CLINICAL TRIAL: NCT06198972
Title: The Effect of Pelvic Proprioceptive Neuromuscular Facilitation (PNF) Exercises on Strength, Balance and Walking Skills in Multiple Sclerosis Patients.
Brief Title: Pelvic Proprioceptive Neuromuscular Facilitation (PNF) Exercises in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZİKKKSU
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: PNF; Pelvic exercise; strength
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): strength exercise training
  Interventions: Other: Strength exercises
- Study Group (Experimental): pnf exercise training
  Interventions: Other: Pelvic Pnf exercises

INTERVENTIONS:
Other: Pelvic Pnf exercises — Exercise Frequency 3 days/week Exercise Intensity 60% of 1 maximum repetition Exercise Duration: 5-minute warm-up 20 minutes (2 sets of 15 repetitions) exercise training 5 min cool down Exercise Type Pelvic patterns
  * Anterior elevation-Posterior depression
  * Anterior depression-Posterior elevation PNF techniques
  * Repetitive stretching
  * Rhythmic stabilization
  Arms: Study Group
Other: Strength exercises — 3 days/week 60% of 1 repetition maximum 5 minute warm up 20 min exercise training 5 min cool down Lower extremity movements
  * Hip flexion
  * Hip extension
  * Hip abduction
  * Hip adduction
  * Knee flexion
  * Knee extension Resistance exercise training
  Arms: Control Group

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune, demyelinating disease that progresses with motor and sensory loss of the central nervous system and causes disability at different levels. Although signs and symptoms vary depending on the location of the lesion, findings such as loss of muscle strength, spasticity, sensory disorders and fatigue cause decreases in walking function in the majority of patients. Loss of muscle strength and fatigue cause loss of mobility, causing individuals with MS to be less physically active than healthy adults in the same age group. As a result, approximately 40% of individuals with MS have walking problems and approximately 70% of them experience a decrease in daily living activities. Literature studies frequently include strengthening exercises for lower extremity muscles in MS patients. However, the results of pelvic pattern exercises, which are the key to lower extremity movements, are not specified. In this study, which is planned in the light of this information, the findings obtained from pelvic PNF exercises will serve to fill this gap in the literature.

DETAILED DESCRIPTION:
According to the data of the Turkish Neurology Association, it is estimated that there are approximately 40,000 MS patients in Turkey. The fact that it is the most common neurological disease in young adults further increases the importance of the need for effective treatment programs.

Exercise training, which aims to improve the functional losses caused by the disease, constitutes a very important part of rehabilitation protocols. For example, while the effects of resistant exercise training have been investigated in athletes and healthy individuals, no definitive results have been obtained regarding correct and effective exercise approaches in MS.

The basic principle of proprioceptive neuromuscular facilitation techniques, defined as facilitating the responses of the neuromuscular mechanism by stimulating the proprioceptors and briefly expressed as PNF, is based on the principle that physiological movements in the human body have rotational and oblique characters and that a greater response can be achieved with movements performed against maximum resistance.

It consists of the pelvis, sacrum, innominate bones (ilium, ischium, pubis) and coccyx. The vertebral column is directly connected to the lower extremities through the sacroiliac joint and is a weight-bearing structure. Pelvic patterns are in harmony with lower extremity patterns. Because the pelvis actually consists of different functional structures and is in relationship with the lower extremities through the hip joint. Pelvic movements and stability are necessary for adequate function of both the trunk and lower extremities. The therapeutic purposes of pelvic patterns are as follows;

* Pelvic movements and stabilization,
* Body stabilization and movements,
* Rotation etc. functional activities,
* To improve lower extremity movements and stabilization Studies conducted on multiple sclerosis patients indicate that walking patterns differ compared to healthy individuals of the same age. Therefore, the main aim of MS rehabilitation is to maintain walking ability and ensure mobility. To this end; Muscle strength, especially proximal muscles, needs to be increased. Also MS; It is a neurological disease that affects the structures responsible for maintaining balance, such as muscle strength and tone, sensory perception, vision and cognition. For this reason, it is reported that balance and gait control are impaired in approximately 80% of MS patients, increasing the number of falls of patients. Because MS disease involves many areas such as the cerebral hemisphere, brainstem and spinal cord, the cause of balance loss may vary from patient to patient. Balance; It is a response formed jointly by visual, sensory, vestibular systems and motor responses. It is complex because of the way systems work together. There is no definitive evidence as to which system is more effective. However, studies have shown that there is a relationship between loss of muscle strength and decreased walking speed and balance problems. It is stated that lower extremity muscle strength is effective on balance because it supports mobility the most and also plays a fundamental role in sensoriomotor functions.

Literature studies frequently include strengthening exercises for lower extremity muscles in MS patients. However, the results of pelvic pattern exercises, which are the key to lower extremity movements, are not specified. In this study, which we planned in the light of this information, the findings obtained from pelvic PNF exercises will serve to fill this gap in the literature.

The hypothesis is that pelvic PNF applications will be superior to lower extremity strengthening exercises in the development of muscle strength, balance and gait in patients with MS who receive 6-week training.

ELIGIBILITY:
Inclusion Criteria:

Consent for the study was obtained;

* Between 18-50 years of age,
* Extended Disability Status Scale (EDSS) score of 4 and below,
* Not in the habit of exercising regularly
* Can walk on the treadmill,
* Not pregnant,
* Not receiving corticosteroid treatment in the last 1 month,
* Fampridine etc. in the last month. not taking medication,
* Patients who have not received Botox treatment in the last 6 months will be included.

Exclusion Criteria:

* Individuals who cannot tolerate the treatment programs and cannot ensure their continuity (2 weeks in a row) will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength: | Baseline and after 6 weeks
  Lower extremity muscle strength will be measured with a digital muscle dynamometer. Lower extremity muscles will be evaluated using a digital dynamometer (Knect). With this device, muscle force values are expressed in Newton (N). Muscle strength will be recorded by making 3 measurements with a digital dynamometer, on the right and left extremities, without allowing the patients to compensate, and the average values will be used.
Figure of 8 walk test | Baseline and after 6 weeks
  It is a standard clinical measurement used to evaluate advanced walking performance required in daily life. In the figure-8 walking test, two cones are placed 1.5 meters apart. The individual stands in the middle of this distance. At the beginning of the test, the child walks around the first cone as fast as he can, then when he reaches the other starting point, this time he walks around the other cone. The elapsed time is recorded. The validity and reliability of the figure-8 walking test was studied in stroke patients and knee prosthesis patients.
12 ıtem walk test | Baseline and after 6 weeks
  It is a 12-item questionnaire that questions the impact of walking on MS. The difficulties experienced by individuals during walking activity in the last 2 weeks are questioned. Each item contains 5 points (1; not at all impressed, 5; completely impressed). Lower scores indicate better gait impairment. It has been reported that the Turkish version of the scale is valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No